CLINICAL TRIAL: NCT04754152
Title: Long-term Effect of θ Burst Magnetic Stimulation on Clinical Symptoms of Alzheimer Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Head, Dept of Neurology & Medical Psychology, Director, Cognitive Neuropsychology Lab, PRC, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHMU-AD-20210103
Record Dates: First submitted 2021-01-30; First posted 2021-02-15 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Repetitive Transcranial Magnetic Stimulation
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TBS Group (Experimental): On the basis of drug treatment, a course of TBS treatment is performed every three months and 4 courses of treatment a year.
  Interventions: Other: θ burst transcranial magnetic stimulation
- Drug Group (Placebo Comparator): Stable doses of cholinesterase inhibitors for the treatment and primary care guidance.Once every 3 months follow-up.
  Interventions: Drug: Pharmacotherapy

INTERVENTIONS:
Other: θ burst transcranial magnetic stimulation — In addition to drug therapy, TBS supplementary therapy was given every 3 months.The TBS parameters were as follows: 3 pulses, 50 Hz bursts given every 200 ms (at 5 Hz), and an intensity of 70% of the resting motor threshold, as measured from the right first dorsal interosseous muscle using a handheld 70 mm figure-of-eight coil. Take a course every 10 weeks .
  Arms: TBS Group
Drug: Pharmacotherapy — Stable doses of cholinesterase inhibitors were given and the patients were followed up every three months.
  Arms: Drug Group

SUMMARY:
This was a randomized, single-blind, parallel, placebo-controlled clinical trial assessing the efficacy of neuronavigational TBS among patients with AD. Fourty late-onset AD were included in the study, all the patients were divided into TBS groups and drug treatment group. Drug intervention group AD patients with drug regimen (donepezil 5mg / d) and primary care guidance, once every three months follow-up. TBS group is treated with TBS (a course of treatment every 3 months); after completing 4 treatments/follow-ups a year, evaluate the changes in MoCA, other clinical symptoms and multi-domain cognition tests, and brain Changes in structure and function.

ELIGIBILITY:
Inclusion Criteria:

* Subject diagnosed with early Alzheimer's disease or related diseases according to NINCDS-ACDRADA criteria.
* Subjects must have a MMSE score between 10 and 27,indicating mild cognitive impairment or dementia
* CDR score ≤ 2
* Subject under treatment by IAChE for at least 3 Weeks.
* psychotropic treatments are tolerated if they were administered and unchanged for at least 3 months

Exclusion Criteria:

* CDR > 2
* Any history or clinical signs of other severe psychiatric illnesses (like major depression,psychosis or obsessive compulsive disorder).

  - Page 5 of 6 [DRAFT] -
* History of head injury,stroke,or other neurologic disease.
* Organic brain defects on T1 or T2 images.
* History of seizures or unexplained loss of consciousness.
* Implanted pacemaker,medication pump,vagal stimulator,deep brain stimulator.
* Family history of medication refractory epilepsy.
* History of substance abuse within the last 6 months.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
changes in Montreal Cognitive Assessment (MoCA) | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  The changes in MoCA will constitute assess response to rTMS the secondary research outcome measure used to.MoCA was developed by Nasreddine et al. based on clinical experience and reference to the MMSE cognitive items and scores, and the final version was finalized in November 2004. We adopted a localized version (Mandarin version#includes 2 alternative versions) in line with the Chinese cultural background.It includes 11 inspection items in 8 cognitive fields, including visual structure skills, executive function, naming, attention and calculation, language, abstract thinking, memory, and orientation. With a total score of 30 or more than 26, it is normal. Anyone who has been education for less than 12 years will need to add one point to his final score. The final score of the higher the better, and we hope the subjects' scores will improve after treatment.

SECONDARY OUTCOMES:
The changes in MMSE(Mini Mental State Examination) | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  The changes in MMSE will constitute the secondary research outcome.The full name of MMSE is mini-mental state examination, and the scale consists of 30 subject, include the following seven aspects: time orientation, place orientation,immediate memory,attention and calculation,delay memory,language, visual space.One point is awarded for each question correctly answered during MMSE evaluation. If subject give the wrong answer or don't know answe he/ she awarded 0 score, scope of scale score of 0 to 30 points. The higher the score, the better. In this study, changes in MMSE scores before and after treatment were used as secondary observations,we hoped that scores would increase after treatment.
HAMD (Hamilton Depression Scale) | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  The changes in HAMD will constitute the secondary research outcome. Hamilton Depression Scale (HAMD) compiled by Hamilton in 1960, is the most common clinical to assess Depression Scale. In this study, 17 versions were selected, and there were 17 questions. The subjects were assessed for their depression in the past week. Each question scored between 0 and 4 points.Higher scores indicate more depressive symptoms. The severity of the disease and the therapeutic effect can be evaluated after treatment. In this study, we hoped that scores would decrease after treatment.
HAMA (Hamilton Anxiety Scale) | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  The changes in HAMA will constitute the secondary research outcome. Hamilton Anxiety Scale (HAMA) was compiled by Hamilton in 1959.It was one of the most commonly used scales in psychiatric clinic, including 14 items. It is often used in clinical diagnosis and degree classification of anxiety disorder. The subjects were assessed for their anxiety in the past week. Each question scored between 0 and 4 points. The higher the score, the more symptoms of anxiety.
  The severity of the disease and the therapeutic effect can be evaluated after treatment. In this study, we hoped that scores would decrease after treatment.
NPI (Neuropsychiatric Inventory) | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  The changes NPI will constitute the secondary research outcome. The Neuropsychology Scale (NPI) evaluates 12 neuropsychiatric disorders which included 10 neuropsychiatric symptoms and 2 autonomic neurological symptoms based on the caregiver's perception of the patient's behavior and the perceived distress. Each item was evaluated for its occurrence frequency (1-4 points) and severity (1-3 points). The frequency and severity were multiplied to obtain the score (0-12 points) of each item.The patient's assessment rating ranges from 0 to 144, and the caregiver's distress rating score is 0 to 60. The lower the score, the lighter the symptoms, and we expect the score to go down after treatment.
ADL( Lawton-Brody Activities of Daily Living) | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  The changes ADL will constitute the secondary research outcome. The ADL evaluates 20 items activities of daily living which included basic life ability and instrument use ability based on the caregiver's perception of the patient's behavior. Each item was evaluated for its severity (1-4 points). The patient's assessment rating ranges from 20 to 80, and the lower the score, the lighter the symptoms, and we expect the score to go down after treatment.
LMT (Logic Memory Test) | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  The changes in LMT will constitute the secondary research outcome.
DST (Digital Span Test; Forward and Backward) | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  The changes in DST will constitute the secondary research outcome. Digital span test (DST) was commonly used to evaluate attention ability and instantaneous memory ability. There are two types of test: forward(0-14) and backward(0-13).In the forward test, the subjects were asked to retell the the digits immediately after hearing it until they could not be repeated correctly.In backward test, the subjects were asked to repeat a set of numbers in reverse order until they could not be repeated correctly. The length of the last set of Numbers correctly repeated by the subjects was the final score, forward and backward are counted separately. The higher the score, the better. In this study, we hoped that scores would increase after treatment.
TMT (Trail Making Test) | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  The changes in TMT will constitute the secondary research outcome. The Trail Making Test (TMT) is divided into two parts, part A and part B. Part A requires the subject to connect 25 Numbers on the paper in sequence, and part B requires the subject to connect 25 Numbers of different colors alternately in sequence. The time it takes for the subject to complete all the Numbers is the subject's final score.In this study, we hoped that scores would decrease after treatment.
JLOT(Judgment of line Judgment of line orientation test orientation test) | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  The changes in JLOT (Judgment of line Judgment of line orientation test orientation test) will constitute assess response to rTMS the secondary research outcome measure.The JLOT test was determined by Benton et al. in 1994.
  There are two versions of H and V. The difference is that the order in which the pictures are presented is different.
  Each version contains 35 images, of which the official test consists of 30 images, and the other 5 images are for the participants to learn. The final score is the correct number of subjects to answer, the full score is 30 points, the higher the score, the better the space perception ability of the subject.We hope the subjects' scores will improve after treatment.
HVOT(Hooper visual organization test Hooper visual organization test) | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  The changes in HVOT(Hooper visual organization test Hooper visual organization test) will constitute assess response to rTMS the secondary research outcome measure.HVOT is a cognitive test used to evaluate the perceived structure of the subject. It consists of 30 items#and each question is 1 point and the total score is 30 points. The final score is the correct number of subjects to answer, the full score is 30 points, the higher the score, the better the space perception ability of the subject.We hope the subjects' scores will improve after treatment.
The Stroop color test | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  The changes in The Stroop color test will constitute assess response to rTMS the secondary research outcome measure.The Stroop color word test was developed by Stroop in 1935 and is used to evaluate the attention function of the subject. The subject is required to correctly read the target color on the stimulus card and record the completion time. The final completion time is the score of the participant. The shorter the time used, the better the performance of the subjects. We expect the participants to spend less time after the real stimulation.
MRI measures | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  Multimodal magnetic resonance data were acquired, including structural phase magnetic resonance and rest state magnetic resonance, to compare the neuroimaging differences between the true and sham stimulation groups before and after stimulation.
Chinese version of the Auditory Verbal Learning Test (AVLT) | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  The changes in AVLT will constitute the secondary research outcome.
Symbol Digit Modalities Test (SDMT) | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  The changes in SDMT will constitute the secondary research outcome.
Verbal Fluency Test-letter and semantic (VFT-L/S). | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  The changes in VFT will constitute the secondary research outcome.
Boston Naming Test (BNT) | baseline; week-2, moth-3, month-6, month-9 and 1-year follow-up
  The changes in BNT will constitute the secondary research outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Cognitive Neuropsychology Lab Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu X, Yan Y, Hu P, Wang L, Wu Y, Wu P, Geng Z, Xiao G, Zhou S, Ji G, Qiu B, Wei L, Tian Y, Liu H, Wang K. Effects of a periodic intermittent theta burst stimulation in Alzheimer's disease. Gen Psychiatr. 2024 Jan 8;37(1):e101106. doi: 10.1136/gpsych-2023-101106. eCollection 2024. PMID 38274292